CLINICAL TRIAL: NCT02917941
Title: A Phase 2, Open-Label, Multicenter Study of Ixazomib Plus Lenalidomide and Dexamethasone in Adult Japanese Patients With Relapsed and/or Refractory Multiple Myeloma
Brief Title: A Study of Ixazomib Plus Lenalidomide and Dexamethasone in Adult Japanese Participants With Relapsed and/or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C16028; U1111-1187-4027 (Other: Universal trial number); JapicCTI-163381 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2016-09-22; First posted 2016-09-28 (Estimated); Results first posted 2020-09-18 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2020-12

CONDITIONS: Relapsed and/or Refractory Multiple Myeloma
MeSH Terms: interventions — ixazomib; Lenalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ixazomib 4 mg + Lenalidomide 25 mg + Dexamethasone 40 mg (Experimental): Ixazomib 4 mg, capsules, orally on Days 1, 8, and 15 plus lenalidomide 25 mg, capsule, orally, once daily on Days 1 through 21 and dexamethasone 40 mg, tablet, orally on Days 1, 8, 15, and 22 of a 28-day cycle up to 32 cycles.
  Interventions: Drug: Ixazomib; Drug: Lenalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Ixazomib — Ixazomib capsules
Drug: Lenalidomide — Lenalidomide capsules
Drug: Dexamethasone — Dexamethasone Tablets

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of ixazomib plus lenalidomide and dexamethasone in Japanese participants with relapsed and/or refractory multiple myeloma (RRMM).

DETAILED DESCRIPTION:
This is a phase 2, open label, single arm, multicenter study to evaluate the efficacy and safety of ixazomib plus lenalidomide and dexamethasone in Japanese participants with relapsed and/or refractory multiple myeloma (MM). The participants population will consist of adult men and women who have a confirmed diagnosis of MM, who have received 1 to 3 prior lines of therapy, and who meet other outlined eligibility criteria. Participants will receive study drug (ixazomib 4.mg) on Days 1, 8, and 15 plus lenalidomide (25 mg) on Days 1 through 21 and dexamethasone (40 mg) on Days 1, 8, 15, and 22 of a 28-day cycle. Participants may continue to receive treatment until progressive disease (PD) or unacceptable toxicity, whichever comes first. Dose modifications may be made based on toxicities. Participant with a low creatinine clearance < 60 mL/min will receive a reduced lenalidomide dose of 10 mg once daily on Days 1 through 21 of a 28-day cycle. The lenalidomide dose may be escalated to 15 mg once daily after 2 cycles if the participant is not responding to treatment and is tolerating the treatment. If renal function normalizes (ie, creatinine clearance >= 60 mL/min) and the participant continues to tolerate this treatment, lenalidomide may then be escalated to 25 mg once daily.

Treatment periods will be defined as 28-day cycles. Participant will be seen at regular treatment cycle intervals while they are participating in the study: four times a treatment cycle for the first 2 cycles, twice a treatment cycle for the 3rd cycle, and then once a treatment cycle for the remainder of their participation in the active treatment and, if applicable, the progression free survival (PFS) and overall survival (OS) follow-up phases of the study.

Response will be assessed by investigator according to the International Myeloma Working Group criteria for all participants every 4 weeks until PD. Central laboratory data will be used for serum M-protein, urine M-protein and serum free light chain. All participants will be followed for survival after progression. Participants will be contacted every 12 weeks until death or termination of the study by the sponsor.

The study will be closed at 24 months from the enrollment of the last participant.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female Japanese participants 20 years of age or older.
2. Multiple myeloma (MM) diagnosed according to standard criteria either currently or at the time of initial diagnosis.

   The initial diagnosis must be symptomatic MM, although the relapsed disease does not need to be symptomatic.
3. Participants must have measurable disease defined by at least 1 of the following 3 measurements based on central laboratory data:

   * Serum M-protein: >=1 g/dL (>= 10 g/L).
   * Urine M-protein: >=200 mg/24 hours.
   * Serum free light chain assay: involved free light chain level >=10 mg/dL (>= 100 mg/L), provided that the serum free light chain ratio is abnormal.
4. Participants with RRMM who have received 1 to 3 prior therapies.

   This participant population includes the following 3 categories of participants:
   * Participants who relapsed from their therapy(s) but were not refractory to any previous therapy.
   * Participants who were refractory to all lines of previous therapy(s) (ie, participants who have never responded to any therapies received).
   * Participants who were relapsed from at least 1 line of therapy AND additionally were refractory to at least 1 line of therapy. For the purposes of this study, refractory MM is defined as PD on therapy or PD within 60 days after the last dose of a given therapy.

   A line of therapy is defined as 1 or more cycles of a planned treatment program. This may consist of 1 or more planned cycles of single-agent therapy or combination therapy, as well as a sequence of treatments administered in a planned manner. For example, a planned treatment approach of induction therapy followed by autologous stem cell transplantation, followed by maintenance is considered 1 line of therapy. Autologous and allogenic transplants are permitted.
5. Participants must meet the following clinical laboratory criteria:

   * Absolute neutrophil count (ANC) >= 1,000/mm3, hemoglobin >= 8 g/dL and platelet count >= 75,000/mm3. Platelet transfusions to help participants meet eligibility criteria are not allowed within 3 days prior to screening.
   * Total bilirubin =< 1.5 x the upper limit of the normal range (ULN).
   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 3 x ULN.
   * Calculated creatinine clearance >= 30 mL/min.
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.
7. Participants who received prior allogenic transplant must have no active graft-versus-host disease (GVHD).
8. Participants who meet the following conditions:

   Female participants who:
   * Are postmenopausal for at least 24 months before the screening visit, OR
   * Are surgically sterile, OR
   * Females of childbearing potential must:

     1. Have a negative pregnancy test with a sensitivity of at least 25 mIU/mL within 10 to 14 days and again within 24 hours prior to starting Cycle 1 of lenalidomide
     2. Agree to practice true abstinence or to begin TWO reliable methods of birth control (1 highly effective method and 1 additional effective method AT THE SAME TIME) for at least 28 days before starting the study treatment through 90 days after the last dose of the study treatment.
     3. Agree to ongoing pregnancy testing
     4. Adhere to the guidelines of the RevMate program

   Male participants, even if surgically sterilized (ie, status postvasectomy), must:
   * Agree to avoid sexual intercourse completely 90 days after the last dose of the study treatment.
   * Agree to practice true abstinence or to practice effective barrier contraception during the entire study treatment period and 90 days after the last dose of the study treatment if their partner is of childbearing potential, even if they have had a successful vasectomy, and
   * Adhere to the guidelines of the RevMate program
9. Thromboembolism prophylaxis is required based on published standard or institutional standard of care.
10. Voluntary written consent must be given before performance of any study-related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the participant at any time without prejudice to future medical care.
11. Participant is willing and able to adhere to the study visit schedule and other protocol requirements.

Exclusion Criteria:

1. Participants who were refractory to lenalidomide or proteasome inhibitor-based therapy at any line.

   Refractory disease is defined as PD on treatment or PD within 60 days after the last dose of a given therapy. Participants who progressed the disease after 60 days from the last dose of a given therapy will be considered relapsed and are eligible for inclusion in the study.

   Participants who were refractory to thalidomide-based therapy are eligible.
2. Female participants who are breast feeding or pregnant.
3. Failure to have fully recovered (ie, =< Grade 1 toxicity) from the effects of prior chemotherapy (except for hair loss) regardless of the interval since the last treatment.
4. Major surgery within 14 days before enrollment.
5. Radiotherapy within 14 days before enrollment.
6. Central nervous system involvement.
7. Infection requiring systemic antibiotic therapy or other serious infection within 14 days before enrollment.
8. Rash or pruritus requiring systemic medication within 14 days before enrollment.
9. Diagnosis of Waldenstrom's macroglobulinemia, polyneuropathy, organomegaly, endocrinopathy, monoclonal gammopathy, and skin changes (POEMS) syndrome, plasma cell leukemia, primary amyloidosis, myelodysplastic syndrome, or myeloproliferative syndrome.
10. Evidence of current uncontrolled cardiovascular conditions, including uncontrolled hypertension, uncontrolled cardiac arrhythmias, symptomatic congestive heart failure, unstable angina, or myocardial infarction within the past 6 months before enrollment.
11. Systemic treatment with strong cytochrome P450, family 3, subfamily A (CYP3A) inducers (rifampicin, carbamazepine, phenytoin), or St. John's wort within 14 days before enrollment.
12. Ongoing or active systemic infection, known human immunodeficiency virus (HIV)- positive, known hepatitis B surface antigen seropositive or known hepatitis C virus (HCV)-RNA positive.

    Participants who have positive hepatitis B core antibody (HBcAb) can be enrolled but must have hepatitis B virus (HBV)-DNA negative. Participants who have positive hepatitis C antibody can be enrolled but must have HCV-RNA negative.
13. Comorbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the participant inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens (eg, peripheral neuropathy that is Grade 1 with pain or Grade 2 or higher of any cause).
14. Psychiatric illness/social situation that would limit compliance with study requirements.
15. Known allergy to any of the study medications, their analogues, or excipients in the various formulations of any agent.
16. Inability to swallow oral medication, inability or unwillingness to comply with the drug administration requirements, or gastrointestinal condition that could interfere with the oral absorption or tolerance of treatment.
17. Diagnosed or treated for another malignancy within 2 years before enrollment or previously diagnosed with another malignancy and have any evidence of residual disease. Participants with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection.
18. Participants who have participated in a clinical trial of ixazomib, or have been treated with ixazomib.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (21):
- Japan (21):
  - Nagoya, Aichi-ken
  - Narita, Chiba
  - Shibukawa, Gunma
  - Fukuyama, Hiroshima
  - Kobe, Hyōgo
  - Ibaraki, Ibaragi
  - Sagamihara, Kanagawa
  - Sendai, Miyagi
  - Ikoma, Nara
  - Sunto-gun, Shizuoka
  - Utsunomiya, Tochigi
  - Bunkyo-ku, Tokyo
  - Koto-ku, Tokyo
  - Shibuya-ku, Tokyo
  - Shinjuku-ku, Tokyo
  - Tachikawa, Tokyo
  - Chiba
  - Fukuoka
  - Niigata
  - Okayama
  - Osaka

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Iida S, Izumi T, Komeno T, Terui Y, Chou T, Ikeda T, Berg D, Fukunaga S, Sugiura K, Sasaki M. A phase 2, open-label, multicenter study of ixazomib plus lenalidomide and dexamethasone in adult Japanese patients with relapsed and/or refractory multiple myeloma. Int J Clin Oncol. 2022 Jan;27(1):224-233. doi: 10.1007/s10147-021-02030-7. Epub 2021 Oct 2. PMID 34599726

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 16 investigative sites in Japan from 01 November 2016 to 31 August 2019.
Pre-assignment Details: Participants with confirmed MM, who received 1-3 lines of prior therapy, received ixazomib 4 mg + lenalidomide and dexamethasone in this study, followed by progression free survival (PFS) and overall survival (OS) follow-up.
Period: Treatment Period
Arm/Group | Ixazomib 4 mg + Lenalidomide 25 mg + Dexamethasone 40 mg
Started | 34
Completed | 10
Not Completed | 24
Not completed — Adverse Event | 11
Not completed — Progressive Disease | 11
Not completed — Reason not Specified | 2
Period: Survival Follow-up Period
Arm/Group | Ixazomib 4 mg + Lenalidomide 25 mg + Dexamethasone 40 mg
Started (Out of 34 Participants, 31 entered the Follow-up Period.) | 31
Completed | 26
Not Completed | 5
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) is defined as all participants who received at least one dose of the study drug during the treatment period.
Arm/Group | Ixazomib 4 mg + Lenalidomide 25 mg + Dexamethasone 40 mg
Number analyzed (Participants) | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.2 (8.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 19
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Not Hispanic or Latino | 34
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian (Japanese) | 34
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 34
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 159.88 (9.738)
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 60.36 (12.444)
Body Surface Area [Mean (Standard Deviation); unit: square meter (m^2)] | 1.632 (0.2076)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Very Good Partial Response (VGPR) or Better Response (Complete Response (CR) + VGPR)
Description: Response was assessed using International Myeloma Working Group (IMWG) Criteria. CR was defined as negative immunofixation in serum and urine and disappearance of any soft tissue plasmacytomas and < 5% plasma cells in bone marrow. VGPR was defined as serum and urine M-protein detectable by immunofixation but not on electrophoresis or 90% or greater reduction in serum M-protein plus urine M-protein level < 100 mg per 24 hours.
Time Frame: Up to approximately 33 months
Population: Response-evaluable analysis set was defined as all full analysis set (FAS) participants with measurable disease at baseline, and at least one postbaseline response assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ixazomib 4 mg + Lenalidomide 25 mg + Dexamethasone 40 mg
Number analyzed (Participants) | 32
percentage of participants | 50.0 [31.9 to 68.1]

2. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the time in months from the date of first study drug administration to the date of first documentation of PD or death from any cause, whichever occurred first. PD required one of the following: increase of ≥ 25% from nadir in: serum M-component (absolute increase ≥ 0.5 g/dl); urine M-component (absolute increase ≥ 200 mg/24 hours); in participants without measurable serum and urine M-protein levels the difference between involved and uninvolved free light chain (FLC) levels (absolute increase > 10 mg/dl); development of new or increase in the size of existing bone lesions or soft tissue plasmacytomas; development of hypercalcemia (corrected serum calcium > 11.5 mg/dl) attributed solely to plasma cell proliferative disease.
Time Frame: Up to approximately 33 months
Population: FAS included all participants who received at least one dose of study drug during the treatment period.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ixazomib 4 mg + Lenalidomide 25 mg + Dexamethasone 40 mg
Number analyzed (Participants) | 34
months | 22.05 [17.28 to NA] — Upper limit of CI was not estimable due to low number of participants with events.

3. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR:percentage of participants with CR including stringent complete response(sCR),VGPR,partial response(PR) per independent review committee(IRC)by IMWG criteria.CR: serum,urine -ve immunofixation; disappearance of soft tissue plasmacytomas,<5%plasma cells in bone marrow(CR in those with only measurable disease by serum FLC levels=normal FLC ratio 0.26 to 1.65+CR criteria).sCR:CR+normal FLC ratio,absence of clonal plasma cells(immunohistochemistry)or 2-to 4-color flow cytometry.VGPR:serum,urine M-protein detectable by immunofixation,not by electrophoresis or ≥90%reduction,<100mg/24hrs(VGPR in those with only measurable disease by serum FLC levels,requires>90%decrease in involved-uninvolved FLC level difference).PR: ≥50%reduction of serum M protein+reduction in 24-hr urinary M protein by≥90%/ to<200mg/24-hr or ≥50%decrease in difference between involved-uninvolved FLC levels/≥50%reduction in bone marrow plasma cells,if≥30%at baseline/≥50%soft tissue plasmacytoma size reduction.
Time Frame: Up to approximately 33 months
Population: Response-evaluable analysis set was defined as all FAS participants with measurable disease at baseline, and at least one postbaseline response assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ixazomib 4 mg + Lenalidomide 25 mg + Dexamethasone 40 mg
Number analyzed (Participants) | 32
percentage of participants | 84.4 [67.2 to 94.7]

4. Secondary Outcome: Duration of Response (DOR)
Description: DOR was measured as time in months from date of first documentation of response, VGPR or better, and ORR (CR+PR (including sCR and VGPR) or better, to date of first documented PD among participants who responded to treatment. Response was assessed by investigator using IMWG Criteria. CR:negative immunofixation in serum and urine and; disappearance of any soft tissue plasmacytomas and;<5% plasma cells in bone marrow. sCR:CR plus normal FLC ratio, absence of clonal plasma cells by immunohistochemistry or 2- to 4-color flow cytometry. VGPR:serum and urine M-protein detectable by immunofixation but not on electrophoresis/≥90% reduction in serum M-protein plus urine M-protein level <100 mg/24 hours. PR:≥50% reduction of serum M protein+reduction in 24-hour urinary M protein by ≥90%/ to <200 mg/24-hour or ≥50% decrease in difference between involved and uninvolved FLC levels/≥50% reduction in bone marrow plasma cells, if ≥30% at baseline/≥50% reduction in size of soft tissue plasmacytomas.
Time Frame: Up to approximately 33 months
Population: FAS included all participants who received at least one dose of study drug during the treatment period. Each responder for VGPR or better, and PR or better in FAS were evaluated in this outcome measure. Responders without documentation of PD were censored at the date of last response assessment that is SD or better.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ixazomib 4 mg + Lenalidomide 25 mg + Dexamethasone 40 mg
Number analyzed (Participants) | 27
months
  VGPR or better: number analyzed (Participants) | 16
  VGPR or better | NA [16.03 to NA] — Median and upper limit of CI was not estimable due to low number of participants.
  ORR | 21.65 [16.03 to NA] — Upper limit of CI was not estimable due to low number of participants.

5. Secondary Outcome: Time to Progression (TTP)
Description: TTP was measured as the time in months from the first dose of study treatment to the date of the first documented PD as assessed using IMWG criteria. PD required one of the following: increase of ≥ 25% from nadir in: serum M-component (absolute increase ≥ 0.5 g/dL); urine M-component (absolute increase ≥ 200 mg/24 hours); in participants without measurable serum and urine M-protein levels the difference between involved and uninvolved FLC levels (absolute increase > 10 mg/dL); development of new or increase in the size of existing bone lesions or soft tissue plasmacytomas; development of hypercalcemia (corrected serum calcium > 11.5 mg/dL) attributed solely to plasma cell proliferative disease.
Time Frame: Up to approximately 33 months
Population: FAS included all participants who received at least one dose of study drug during the treatment period.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ixazomib 4 mg + Lenalidomide 25 mg + Dexamethasone 40 mg
Number analyzed (Participants) | 34
months | 22.57 [17.51 to NA] — Upper limit of CI was not estimable due to low number of participants with events.

6. Secondary Outcome: Number of Participants With One or More Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is any unfavorable or unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product whether or not it was related to the medicinal product. A TEAE is defined as any AE that occurred after administration of the first dose of any study drug through 30 days after the last dose of any study drug.
Time Frame: Up to approximately 33 months
Population: Safety analysis set included all participants who received at least one dose of study drug during the treatment period.
Measure: Count of Participants; unit: Participants
Arm/Group | Ixazomib 4 mg + Lenalidomide 25 mg + Dexamethasone 40 mg
Number analyzed (Participants) | 34
Participants | 34

7. Secondary Outcome: Number of Participants With NCI CTCAE Grade 3 or Higher TEAEs Related Laboratory Parameters
Description: Laboratory parameters included chemistry and hematology. An AE is any unfavorable or unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product whether or not it was related to the medicinal product. A TEAE is defined as any AE that occurred after administration of the first dose of any study drug through 30 days after the last dose of any study drug. An AE was graded as per NCI CTCAE.
Time Frame: Up to approximately 33 months
Population: Safety analysis set included all participants who received at least one dose of study drug during the treatment period. Number analyzed is the number of participants with data available for analyses for the specific category.
Measure: Count of Participants; unit: Participants
Arm/Group | Ixazomib 4 mg + Lenalidomide 25 mg + Dexamethasone 40 mg
Number analyzed (Participants) | 34
Participants
  Platelet count decreased | 7
  Neutrophil count decreased | 6
  White blood cell count decreased | 3
  Lymphocyte count decreased | 1
  Alanine aminotransferase increased | 1
  Aspartate aminotransferase increased | 1
  Lipase increased: number analyzed (Participants) | 33
  Lipase increased | 1
  Blood creatine phosphokinase increased | 1

8. Secondary Outcome: Number of Participants With NCI CTCAE Grade 3 or Higher TEAEs Related to Vital Signs
Description: Vital signs included temperature, blood pressure, heart rate, and respiratory rate. An AE is any unfavorable or unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product whether or not it was related to the medicinal product. A TEAE is defined as any AE that occurred after administration of the first dose of any study drug through 30 days after the last dose of any study drug. An AE was graded as per NCI CTCAE.
Time Frame: Up to approximately 33 months
Population: Safety analysis set included all participants who received at least one dose of study drug during the treatment period.
Measure: Count of Participants; unit: Participants
Arm/Group | Ixazomib 4 mg + Lenalidomide 25 mg + Dexamethasone 40 mg
Number analyzed (Participants) | 34
Participants
  Hypertension | 1
  Hypotension | 1

9. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of first study drug administration to the date of death.
Time Frame: Up to approximately 33 months
Population: FAS included all participants who received at least one dose of study drug during the treatment period. Participants without documentation of death at the time of the analysis were censored at the date when they were last known to be alive.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ixazomib 4 mg + Lenalidomide 25 mg + Dexamethasone 40 mg
Number analyzed (Participants) | 34
months | NA [30.85 to NA] — Median and upper limit of overall survival was not estimable due to low number of participants with events.

ADVERSE EVENTS:
Time Frame: Up to approximately 33 months
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Ixazomib 4 mg + Lenalidomide 25 mg + Dexamethasone 40 mg
All-Cause Mortality (participants affected / at risk) | 3/34
Serious Adverse Events (participants affected / at risk) | 12/34
Other Adverse Events (participants affected / at risk) | 34/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ixazomib 4 mg + Lenalidomide 25 mg + Dexamethasone 40 mg (N=34)
Pneumonia (Infections and infestations) | 3
Cellulitis (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Inguinal hernia (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Fall (Injury, poisoning and procedural complications) | 2
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1
Platelet count decreased (Investigations) | 1
Blood creatine phosphokinase increased (Investigations) | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1
Hypotension (Vascular disorders) | 1
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 1
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant neoplasm of unknown primary site (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1
Subarachnoid haemorrhage (Nervous system disorders) | 1
Loss of consciousness (Nervous system disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Lung neoplasm malignant (Respiratory, thoracic and mediastinal disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Sebaceous naevus (Congenital, familial and genetic disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ixazomib 4 mg + Lenalidomide 25 mg + Dexamethasone 40 mg (N=34)
Constipation (Gastrointestinal disorders) | 17
Diarrhoea (Gastrointestinal disorders) | 14
Nausea (Gastrointestinal disorders) | 10
Vomiting (Gastrointestinal disorders) | 5
Abdominal distension (Gastrointestinal disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 3
Dental caries (Gastrointestinal disorders) | 5
Gastritis (Gastrointestinal disorders) | 2
Haemorrhoids (Gastrointestinal disorders) | 2
Stomatitis (Gastrointestinal disorders) | 4
Upper respiratory tract infection (Infections and infestations) | 16
Nasopharyngitis (Infections and infestations) | 11
Bronchitis (Infections and infestations) | 6
Pharyngitis (Infections and infestations) | 5
Influenza (Infections and infestations) | 7
Conjunctivitis (Infections and infestations) | 3
Cystitis (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 2
Rash (Skin and subcutaneous tissue disorders) | 12
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5
Urticaria (Skin and subcutaneous tissue disorders) | 4
Dry skin (Skin and subcutaneous tissue disorders) | 4
Erythema multiforme (Skin and subcutaneous tissue disorders) | 3
Asteatosis (Skin and subcutaneous tissue disorders) | 2
Malaise (General disorders) | 5
Oedema peripheral (General disorders) | 5
Pyrexia (General disorders) | 4
Face oedema (General disorders) | 2
Fatigue (General disorders) | 2
Platelet count decreased (Investigations) | 9
Neutrophil count decreased (Investigations) | 6
White blood cell count decreased (Investigations) | 3
Aspartate aminotransferase increased (Investigations) | 2
Weight decreased (Investigations) | 2
Dysgeusia (Nervous system disorders) | 7
Peripheral sensory neuropathy (Nervous system disorders) | 7
Headache (Nervous system disorders) | 3
Dizziness (Nervous system disorders) | 2
Neuralgia (Nervous system disorders) | 3
Chillblains (Injury, poisoning and procedural complications) | 7
Fall (Injury, poisoning and procedural complications) | 5
Arthropod bite (Injury, poisoning and procedural complications) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4
Neutropenia (Blood and lymphatic system disorders) | 7
Thrombocytopenia (Blood and lymphatic system disorders) | 4
Anaemia (Blood and lymphatic system disorders) | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 4
Decreased appetite (Metabolism and nutrition disorders) | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4
Insomnia (Psychiatric disorders) | 2
Renal impairment (Renal and urinary disorders) | 2
Periodontal disease (Gastrointestinal disorders) | 2
Contusion (Injury, poisoning and procedural complications) | 2
Tooth fracture (Injury, poisoning and procedural complications) | 2
Hyperlipidaemia (Metabolism and nutrition disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2016-11-25): https://cdn.clinicaltrials.gov/large-docs/41/NCT02917941/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-19): https://cdn.clinicaltrials.gov/large-docs/41/NCT02917941/SAP_001.pdf